CLINICAL TRIAL: NCT00865306
Title: Early Intervention for Children at Risk for Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Dina Hirshfeld-Becker, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000P000305; K08MH001538 (NIH)
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Results first posted 2010-10-13 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-09

CONDITIONS: Anxiety Disorder
Keywords: Cognitive behavioral therapy; Anxiety; Preschoolers; Young Children; Parents; At-risk; Behavioral Inhibition
MeSH Terms: conditions — Anxiety Disorders | interventions — Coping Skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active CBT (Experimental): Seven parent-only and 8-13 child-only sessions focusing on CBT for anxiety disorders using the "Being Brave" protocol.
  Interventions: Behavioral: "Being Brave: A Program for Coping with Anxiety for Young Children and Their Parents."
- No intervention (wait-list controls) (No Intervention): Control children received no intervention.

INTERVENTIONS:
Behavioral: "Being Brave: A Program for Coping with Anxiety for Young Children and Their Parents." — This is a cognitive-behavioral intervention modeled loosely after Kendall's "Coping Cat," which includes 7 parent-only sessions and 8-13 child-only sessions. It focuses on helping parents learn strategies for coaching their child in coping with anxiety, and on teaching the child coping skills and carrying out exposure exercises in session and in parent-child homework assignments.
  Arms: Active CBT

SUMMARY:
The aim of this study was to develop and pilot a cognitive-behavioral therapy (CBT) parent-child intervention for 4-7-year-old children at risk for anxiety disorders. The 20-session intervention was first piloted openly in 9 children (between 3/10/98 and 1/1/2001). The intervention was then tested in 65 children in a randomized controlled trial versus a monitoring-only wait-list control condition. Children had to either have an anxiety disorder, behavioral inhibition, or be the offspring of a parent with an anxiety disorder who had elevated symptoms of anxiety. In practice all children but one had at least one anxiety disorder at baseline. Children were blocked on presence or absence of parental anxiety disorder and randomized to the intervention or to a no-intervention wait-list control group. The intervention consisted of 6 parent-only sessions, 8-13 child-parent sessions, and a final parent session. Post-trial assessments were conducted at six months, and at one-year follow-up. The hypotheses were that the children assigned to the intervention group would show significantly better improvement (measured via Clinician Global Impression-Anxiety Improvement scale and absence of anxiety disorders) than children assigned to the wait-list condition.

ELIGIBILITY:
Inclusion Criteria:

* The child is at risk for anxiety disorders, as indicated by at least one of the following:
* the child has behavioral inhibition (as determined by observed behavioral assessment);
* the child meets criteria for a DSM-IV or IIIR anxiety disorder (as determined by Kiddie-Schedule for Affective Disorders and Schizophrenia, Epidemiologic Version [K-SADS-E] with the mother); or
* the child has both a parent with lifetime history of anxiety disorder (as determined by direct Structured Clinical Interview for DSM-IV [SCID-IV] with both parents) and the child has anxious symptomatology, as indicated by Child Behavior Checklist [CBCL] scale scores (T-scores) on Anxious/Depressed or Withdrawn of 55 or higher.
* The child is between the ages of 4 and 7 years
* The child and parent(s) have a working command of English

Exclusion Criteria:

* Psychosis in parent or child
* Suicidality in parent or child
* Current alcohol or substance abuse in a parent
* Mental retardation or pervasive developmental disorder in parent or child
* Child in current psychiatric treatment
* Child judged too uncooperative or distractible to take part in intervention
* (In the controlled trial): Child judged clinically unable to wait six months for treatment. The following criteria are used in determining whether the child can wait for 6 months before receiving treatment:
* Suicidal Ideation
* Serious impairment in eating or sleeping habits
* Severe social isolation
* Severe impairment in school functioning or attendance
* Severe symptoms of obsessive-compulsive disorder (OCD)
* Clinical judgment based on the child's overall severity of symptoms and family functioning.
* All judgments of severity of symptoms/impairment are based on a clinician review of the Kiddie-SADS-E and a clinical evaluation with the family.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 1998-03; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dina Hirshfeld-Becker, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States

REFERENCES:
- [Result] Hirshfeld-Becker DR, Masek B, Henin A, Blakely LR, Pollock-Wurman RA, McQuade J, DePetrillo L, Briesch J, Ollendick TH, Rosenbaum JF, Biederman J. Cognitive behavioral therapy for 4- to 7-year-old children with anxiety disorders: a randomized clinical trial. J Consult Clin Psychol. 2010 Aug;78(4):498-510. doi: 10.1037/a0019055. PMID 20658807

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment for the controlled trial occurred between February 2001 and January 2004. Children were recruited from the outpatient child psychiatry clinic at a general hospital, as well as through print ads in local newspapers and parent magazines, email advertisements to hospital employees, and posters at local pediatrics practices.
Pre-assignment Details: We screened 103 children for the controlled trial, to enroll our target goal of 60-65 children. Of these 14 were ineligible (3 did not meet inclusion criteria, and 9 met exclusion criteria). Another 13 withdrew prior to completing baseline assessments, and 11 who did not complete baseline assessments were lost to follow-up. Thus 65 were enrolled.
Groups:
- Active CBT: This was parent-child CBT, administered to families individually over 6 months, and including six 1-hour parent-only sessions, followed by 8-13 1-hour child-parent sessions, and one final 1-hour parent-only session.
- No Intervention (Wait-list Controls): This was a 6-month wait-list control condition in which children received no intervention. After participating in the control condition, families who wanted it were offered the opportunity to receive the CBT intervention.
Period: Controlled Trial
Arm/Group | Active CBT | No Intervention (Wait-list Controls)
Started | 34 (35 assigned to CBT. One child in trial had 0 anxiety disorders, so we excluded her from analysis.) | 30
Completed | 29 | 28
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Difficulty commuting | 2 | 0
Not completed — Improved btw baseline and first session | 1 | 0
Not completed — Sought treatment for conduct disorder | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: One-Year Follow-Up
Arm/Group | Active CBT | No Intervention (Wait-list Controls)
Started | 29 | 15 (Only controls who opted for CBT after the waitlist (n=17) were included. 2 were lost (15 included).)
Completed | 29 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active CBT | No Intervention (Wait-list Controls) | Total
Number analyzed (Participants) | 34 | 30 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 34 | 30 | 64
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] — The mean age of the children was 5.4 years (SD 1.0). This value did not differ between groups.
  years | 5.4 (1.0) | 5.4 (1.0) | 5.4 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 17 | 13 | 30
Region of Enrollment [Number; unit: participants]
  United States | 34 | 30 | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders Based on Clinician Global Impression-Anxiety Improvement
Description: Clinicians blind to treatment assignment rated the child's global improvement on anxiety, using the Clinician Global Impression-Anxiety Improvement scale (CGI-Anxiety, best value 1, worst value 7). Responders were considered those with "very much" or "much" improvement (CGI-Anxiety scores of 1 or 2)
Time Frame: Post-Treatment (6-months from baseline)
Measure: Number; unit: Participants
Arm/Group | Active CBT | No Intervention (Wait-list Controls)
Number analyzed (Participants) | 34 | 30
Participants | 20 | 9
Statistical Analysis 1: Comparison: Active CBT vs No Intervention (Wait-list Controls); Test type: Superiority or Other; p < .05, Chi-squared

2. Other Pre Specified Outcome: Number of Children Free of Anxiety Disorders
Description: Number of children free of anxiety disorders, as assessed by clinicians blind to treatment condition.
Time Frame: Post-Treatment (6-months from baseline)
Measure: Number; unit: Participants
Arm/Group | Active CBT | No Intervention (Wait-list Controls)
Number analyzed (Participants) | 34 | 30
Participants | 17 | 5
Statistical Analysis 1: Comparison: Active CBT vs No Intervention (Wait-list Controls); Test type: Superiority or Other; p < .01, Chi-squared

3. Other Pre Specified Outcome: Number of Responders Using Clinical Global Impression-Anxiety Improvement at 1-Year Follow-Up
Description: Clinicians rated improvement on anxiety since baseline using the Clinical Global Impression-Anxiety Improvement scale (Best 1, Worst 7), with children considered responders if they were rated "1, very much improved" or "2, much improved." Note that rates for controls are for controls who were subsequently treated with CBT (after completing the wait-list control condition).
Time Frame: 1-Year Follow-Up
Population: We tabulated the number of children that were "much" or "very much" improved on anxiety since baseline. Note that the controls who were followed up at one-year were those who subsequently received CBT (after participating in the wait-list condition). Therefore the "No intervention (wait-list controls)" followed up here had actually received CBT.
Measure: Number; unit: Participants
Arm/Group | Active CBT | No Intervention (Wait-list Controls)
Number analyzed (Participants) | 29 | 15
Participants | 24 | 11

ADVERSE EVENTS:
Arm/Group | Active CBT | No Intervention (Wait-list Controls)
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/30
Other Adverse Events (participants affected / at risk) | 0/34 | 0/30

LIMITATIONS AND CAVEATS:
Wait-list control condition Use of parent report in diagnostic interviews (necessary in this young age range) Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No